CLINICAL TRIAL: NCT06162975
Title: The Surveillance (Non-interventional, Observational) Clinical Study of Rickettsiosis Caused by a New Genotype of Rickettsia in the Altai Republic, Russian Federation
Brief Title: The Surveillance Clinical Study of Rickettsiosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Other Study IDs: 01-RICK-2023
Record Dates: First submitted 2023-11-28; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Rickettsiosis
MeSH Terms: conditions — Rickettsia Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this surveillance (non-interventional) clinical study is to genotype the causative agents of rickettsiosis in biological samples of patients from the Altai Republic, Russian Federation. This is a solely observational study in the patients with diagnosed or suspected tick-borne rickettsioses, with no intervention to the routine treatment and diagnostic process. During the study the medical history, diseases progress and symptoms, as well as treatments are being registered in individual case report forms. The rests of the samples used for standard diagnostics (plasma, or serum, and/or swabs of the tick bite site) are being collected and afterwards will be analyzed for a new rickettsia type. These data will be compared to the medical history and symptoms of the patients in order to identify clinical pattern specific for the new rickettsia type. Informed consents from all patients or their legal representatives are being collecting. The study was approved by the local ethical committee.

ELIGIBILITY:
Inclusion Criteria:

* Written patient's informed concent for study participation;
* Male and female patients of any age with diagnosed or suspected tick-born rickettsioses.

Exclusion Criteria:

- Unwillingness to participate in the study by any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients of any age with diagnosed or suspected tick-born rickettsioses.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Genotype the causative agents of rickettsiosis | up to 4 weeks
  Genotype the causative agents of rickettsiosis in biological samples (blood and swab) of patients from the Altai Republic, Russian Federation

CONTACTS AND LOCATIONS:
Locations (1):
- Altai Republic Center for HIV prophylaxis and treatment, Gorno-Altaysk, Altai Republic, Russia

IPD SHARING:
Plan to Share IPD: No